CLINICAL TRIAL: NCT05696288
Title: Conventional Oxygen Therapy Versus Continuous Transnasal High Flow Oxygen Therapy for Head and Neck Diagnostic Panendoscopy Under General Anesthesia in Spontaneous Ventilation
Acronym: OPTINOSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022/16
Record Dates: First submitted 2023-01-11; First posted 2023-01-25 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: To compare the incidence of oxygen desaturation in patients ventilated with the Optiflow™ system to that of patients treated according to the standard technique.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: investigational device (Respiratory Gas Delivery System) (Experimental): Patients ventilated with the Optiflow™ system, a nasal high flow oxygenation system (NHFO) while undergoing a panendoscopy
  Interventions: Procedure: Respiratory Gas Delivery System
- Arm B: standard nasal oxygenation device (Active Comparator): Patients ventilated according to the standard technique while undergoing a panendoscopy
  Interventions: Procedure: Respiratory Gas Delivery System

INTERVENTIONS:
Procedure: Respiratory Gas Delivery System — Oxygen therapy during general anesthesia for ENT panendoscopy

SUMMARY:
The high-flow oxygen therapy system, also called the THRIVE (Transnasal Humidified Rapid-Insufflation Ventilatory Exchange) system, appears to provide better patient safety than conventional techniques.

Panendoscopy is a very common diagnostic procedure in ENT surgery. The general anesthesia during the diagnostic panendoscopy is a good representation of the induction stage. Indeed, the procedure of preoxygenation preceding anesthetic induction and direct laryngoscopy corresponds to the airway management that is an integral part of each general anesthesia. This is why researchers are studying it in particular to improve patient safety during difficult intubations. The paradox is that there is no consensus on the anesthetic strategy for this procedure that counts four main methods for the airway management of patients requiring an ENT panendoscopy. In our center, the investigators use, in most situations, a variant of spontaneous ventilation described by Y. Jacquet et al., with the difference that the investigators use a transglottic oxygenation probe during the procedure. During laryngoscopy, the operator positions a naso-tracheal tube after local anesthesia of the vocal cords. The oxygen flow is reduced to 3 L/min before the exploration procedure. The arrival in operating theaters of the Optiflow™ system, developed by the New Zealand Company Fisher & Paykel Healthcare, has led to a rethinking of the way oxygen is delivered. This device allows the administration of a flow rate of up to 70 L/min while delivering heated gases.

DETAILED DESCRIPTION:
This device allows the administration of a flow rate of up to 70 L/min while delivering heated gases. The benefit of Optiflow™ no longer needs to be demonstrated for certain intensive care patients. In the field of Anesthesia, the number of publications raised up since the increase in the non-hypoxemic apnea time during general anesthesia is never equaled by other methods.

What is known is that panendoscopy under general anesthesia in spontaneous ventilation is not unanimously accepted due to a higher risk regarding the time allowed for apnea, and laryngospasm complications. High-flow oxygen delivery provide a longer safe apnea time for patient safety. The aim of this investigation is to prove that high-flow oxygen therapy improves patient safety during general anesthesia for ENT panendoscopy. This should allow answering the question: shouldn't very high flow oxygenation be systematically offered for this procedure? Currently, there is no consensus as to the anaesthetic strategy for this procedure, if our hypothesis is verified; the Optiflow™ system could become de gold standard of the management of the upper airway during the ENT procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from a head and neck cancer, most often tumor of the bucco-pharyngo-laryngeal cavities, having to carry out a diagnostic HN panendoscopy;
* Patient over 18 years of age;
* ASA < 4;
* BMI ≤ 45;
* Patient willing and able to provide written informed consent for the trial;;
* Patient affiliated with a health insurance system.

Exclusion Criteria:

* Patient with a contraindication to the Optiflow™ system as defined in the manufacturer's brochure;
* Patient with a tumor obstructing more than 80% of the glottic lumen;
* Patient with impossible intubation criteria:

  * Mallampati 4 and mouth opening less than 20 mm
  * Retrognathia
* Patient with:

  * A known intracranial pathology;
  * Documented pulmonary hypertension;
  * Uncontrolled epilepsy;
  * Uncontrolled heart rhythm disorder;
  * Pulmonary pathology with hypoxemia: Spo2 <92% in ambient air;
* Patient at high risk of a full stomach evaluated by the anesthetist;
* ASA ≥ 4
* Morbid obesity with BMI> 45;
* Obstructive upper airway tumor with functional impact;
* Known contraindication to propofol or alfentanil;
* Panendoscopy procedure to be combined with an oesogastro-duodenal fibroscopy;
* Vulnerable persons as defined by articles 64 and 68 of Regulation (EU) 2017/745 of the European Parliament and of the Council of 5 April 2017 on medical devices :

  * In the case of incapacitated subjects who have not given, or have not refused to give, informed consent before the onset of their incapacity, a clinical investigation may be conducted only where, in addition to the conditions set out in Article 62(4)
  * Pregnant or breast-feeding women who do not fall under the provisions of Article 66
  * Adults subject to a legal protection order or unable to give their consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Incidence of arterial desaturation | 1 day, during the procédure
  The O2 saturation defined as SpO2 <95% will be collected each time it reaches 94% or less

SECONDARY OUTCOMES:
Measure the non-hypoxemic apnea time | 1 day, during the procédure
  Non-hypoxemic apnea time will be measured as soon as the SpO2 parameter is between 100 and 95%
Incidence of the use of manual ventilation | 1 day, during the procedure
  Interruption of the surgical procedure for use of manual ventilation with a facemask will be recorded.
Incidence of the use of tracheal intubation | 1 day, during the procedure
  Conversion from the OHD oxygenation technique to the standard technique will be recorded
Incidence of the use of neuromuscular blocking drugs | 1 day, during the procedure
  The use of neuromuscular blocking drugs will be recorded
Incidence of emergency tracheostomy | 1 day, during the procedure
  The performance of an emergency tracheostomy will be recorded
Incidence of complications in SSPI and the complication rate on D1 after the panendoscopy procedure | Through study completion, up to 2 days
  Occurrence of complications in SSPI and on D1 after the panendoscopy procedure will be recorded. Complication in SSPI is define as prolonged desaturation requiring a supply of ventilation whatever the modalities, symptomatic hypercapnia or cardiovascular complications.
Correlation between sedation dose and duration of non-hypoxemic apnea | 1 day, during the procedure
  Correlation between the dose of sedation and the duration of non-hypoxemic apnea will be evaluated using Spearman's R coefficient
Evaluation of the technique fluctuation | 1 day, during the procedure
  Hypoxic desaturation will be reported by acts and by technique
Operator satisfaction | 1 day, after the procedure
  Operator's satisfaction will be noted at the end of each procedure using a visual analogic scale from 1 to 6
Patient satisfaction | up to 2 days
  Patient satisfaction will be recorded using a scale from 1 to 6

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Henri KOULMANN, MD, Principal Investigator — Centre Antoine Lacassagne
Locations (1):
- Centre Antoine Lacassagne, Nice, France